CLINICAL TRIAL: NCT00372099
Title: Evaluation of the Effects of Salmon Calcitonin Nasal Spray Compared to Placebo on Bone Microarchitecture Measured by High Resolution Peripheral Micro- Computed-tomography Over 2 Years in Postmenopausal Women (a Pilot Study)
Brief Title: Bone Microstructure in Nasal Salmon Calcitonin Treated Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rene Rizzoli (Other)
Responsible Party: Sponsor-Investigator, Rene Rizzoli, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-262/Psy 05-038; CSMC051ACH01
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Postmenopause
Keywords: Postmenopausal women; bone microarchitecture; peripheral quantitative micro-CT; salmon calcitonin
MeSH Terms: interventions — salmon calcitonin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Salmon calcitonin — nasal salmon calcitonin 200UI/day during 2 years

SUMMARY:
Calcitonin has been used for many years for treating osteoporosis in postmenopausal women. Recent data from the 2 years placebo-controlled QUEST study have shown a preservation of microarchitecture as measured by high resolution MRI in postmenopausal women with prevalent vertebral fractures at baseline.This pilot study should provide additional new insights in the mode of action of nasal calcitonin, on structural changes as measured by high resolution peripheral CT, and on the comparison between weight bearing and non weight bearing bones in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Women between age 45-70
* Natural or surgical menopause ≥ 1 year
* T-Score between 0.0 and -2.49 (spine or proximal femur - total or femoral neck measured by DXA)

Exclusion Criteria:

* Osteoporosis (T-score ≤ -2.5 in spine or proximal femur - total or femoral neck, measured by DXA)
* Severe vertebral fracture, as identified by screening DXA assessment
* Any history of metabolic disease, which could affect bone metabolism: hyperparathyroidism, osteogenesis imperfecta, Paget's disease, osteomalacia
* Thyroid disease (if receiving thyroid hormone replacement, the patients must be euthyroid, and on a stable dose of thyroid hormone)
* Impaired renal function (estimated GFR<30 ml/min)
* History of previous or active malignancy of any organ system, treated or not treated within the past 5 years.
* History of corticosteroids treatments during 6 months or more, daily dosage >5 mg .
* BMI < 18 or >30.
* Treatments with estrogens, SERMs, tibolone, calcitonin, strontium ranelate, teriparatide or PTH, oral or iv bisphosphonates in the previous year.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-01; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Bone micro-architecture evaluated by high resolution p-QCT | 24 months

SECONDARY OUTCOMES:
Bone turn-over markers | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: René Rizzoli, Professor, Principal Investigator — Department of Rehabilitation and Geriatrics, University Hospital of Geneva

REFERENCES:
- [Derived] Richert L, Uebelhart B, Engelhardt M, Azria M, Rizzoli R. A randomized double-blind placebo-controlled trial to investigate the effects of nasal calcitonin on bone microarchitecture measured by high-resolution peripheral quantitative computerized tomography in postmenopausal women - study protocol. Trials. 2008 Apr 13;9:19. doi: 10.1186/1745-6215-9-19. PMID 18405390